CLINICAL TRIAL: NCT03114384
Title: Patient-ventilator Asynchrony During Noninvasive Ventilation Assessed Using Diaphragm Ultrasonography
Acronym: ADULT
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Centre Hospitalier Saint Joseph Saint Luc de Lyon (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: 2017-A00346-47
Record Dates: First submitted 2017-04-10; First posted 2017-04-14 (Actual); Last update posted 2017-04-14 (Actual); Status verified 2017-04

CONDITIONS: Diaphragm; Ultrasonography
MeSH Terms: interventions — Facility Design and Construction

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Healthy volunteers (Experimental)
  Interventions: Other: Creation and detection of patient-respirator asynchronies

INTERVENTIONS:
Other: Creation and detection of patient-respirator asynchronies — The provocation of leaks on the Ventilation circuit and expiratory trigger modulation will generate a number of asynchronies between the subject and the respirator

SUMMARY:
Fifteen healthy subjects under non-invasive ventilation will be have a recording of surface electromyogram, measurements of airway flows and pressures as well as a continuous ultrasound. The provocation of leaks on the Ventilation circuit and expiratory trigger modulation will generate a number of asynchronies between the subject and the respirator.

These records will help to assess the agreement between the detection of asynchronies using electromyography of the respiratory muscles (technique of reference) and the diaphragmatic echography. We will also compare the respective performance of two techniques of diaphragmatic exploration (excursion and thickening of the diaphragm). A sensitivity of Ultrasound technique of at least 90% will be interpreted as a satisfactory index of concordance.

ELIGIBILITY:
Inclusion Criteria:

* Healthy volunteer (male or female)
* Free and Informed Consent

Exclusion Criteria:

* Known pregnancy, parturient or nursing mother
* Minor under 18 years of age
* Major incapable
* Non-affiliation to the social security scheme
* Any history of respiratory pathology

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 15 (Estimated)
Dates: Start 2017-04-14 (Estimated); Primary Completion 2017-07-30 (Estimated); Study Completion 2017-07-30 (Estimated)

PRIMARY OUTCOMES:
Asynchronies detection with diaphragm ultrasonography | thirty minutes
  Evaluation of the agreement between asynchronous subject-ventilator detection using diaphragm ultrasonography and detecting the same events in using the electromyogram of the respiratory muscles (as a reference technique.

CONTACTS AND LOCATIONS:
Locations (1):
- Groupe Hospitalier Henri Mondor, Créteil, France

IPD SHARING:
Plan to Share IPD: No